CLINICAL TRIAL: NCT06074367
Title: Post Operative Atril Fibrillation : The Impact of Oral Vitamin C in Reducing the Risk in Egyptian CABG Patients
Brief Title: The Impact of Oral Vitamin C in Prevention for Post Operative Atrial Fibrillation (POAF) in Coronary Artery Bypass Surgery (CABG) Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Sahar Mohamed Hesham, principle investigator, Helwan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Vitamin C in POAF prevention
Record Dates: First submitted 2023-08-25; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Post Operative Atrial Fibrillation
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The study was double blinded were Participant (patients), Care Provider (nurses, cardiac surgeons, and ICU physicians) were blinded but the outcome assessors (clinical pharmacist) who collect data were not blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP 1 (2g Vitamin C ) (Experimental)
  Interventions: Drug: Vitamin C 500 MG Oral Capsule(High dose 2g daily)
- GROUP 2 (1g Vitamin C ) (Experimental)
  Interventions: Drug: Vitamin C 500 MG Oral Capsule(Low-dose 1g daily)
- Control group (Placebo Comparator)
  Interventions: Drug: placebo capsules

INTERVENTIONS:
Drug: Vitamin C 500 MG Oral Capsule(High dose 2g daily) — A sixty CABG patients commenced on maximum tolerated dose of b-blocker, statins & vitamin C 500 mg (2 g-daily in 4 divided doses) started one day before operation till the end of hospital stay or development of post operative atrial fibrillation
  Arms: GROUP 1 (2g Vitamin C )
Drug: Vitamin C 500 MG Oral Capsule(Low-dose 1g daily) — A sixty CABG patients commenced on maximum tolerated dose of b-blocker, statins, vitamin C 500 mg (1 g-daily in 2 divided doses) and also received 2 capsules containing starch to be completely equivalent in frequency to the other groups. the intervention started one day before operation till the end of hospital stay or development of post operative atrial fibrillation.
  Arms: GROUP 2 (1g Vitamin C )
Drug: placebo capsules — A sixty CABG Patients commenced on maximum tolerated dose of b-blocker, statins and placebo capsules containing starch mimic vitamin C capsules was taken every 6 hrs. The placebo capsules were prepared in the same shape and size as the original ones manufactured by the same pharmaceutical company. the intervention started one day before operation till the end of hospital stay or development of post operative atrial fibrillation.
  Arms: Control group

SUMMARY:
Post operative atrial fibrillation (POAF) is one of the most common complications that takes place worldwide after coronary artery bypass surgeries (CABG). Many studies suggest using vitamin C as an additional treatment alongside standard therapies, such as statins and β-blockers, to reduce the risk of postoperative atrial fibrillation (POAF) in patients undergoing (CABG). Supplemental therapy with vitamin C may provide a more robust preventive effect against POAF compared to using statins and β-blockers due to its strong antioxidant effect. This implies that vitamin C can enhance the effectiveness of those medications used for POAF prevention by decreasing oxidative stress induced by the surgery.

There are conflicting data on whether or not vitamin C as an antioxidant has a protective effect against postoperative atrial fibrillation and has a significant role in shortening length of ICU and hospital stay . Even in those studies that show positive relationship of vitamin C in AF prevention, there is a diversity in the dosing regimen of vitamin C used among those previous studies.

To the best of our knowledge, most researches were conducted predominantly within a single geographic region, such as Iran, this raises the concerns about the potential bias and limits our ability to apply the findings to a broader global population.

Here, the investigators aimed to evaluate the effectiveness of vitamin C supplementation and to figure out which dose of vitamin C will prevent post-operative AF and decrease complications such as hospital stay, pneumonia and surgical site infection among older Egyptian adults.

ELIGIBILITY:
Inclusion criteria:

* Patients who underwent elective isolated on-pump coronary artery bypass surgery
* Age: 50 to 70 years
* No history of Coronary artery by pass surgery
* Taking maximum tolerated beta-blocker before and after surgery
* Normal left atrium and left ventricle dimensions

Exclusion Criteria:

* preoperative history of Atrial fibrilliation
* permanent pacemaker or significant bradycardia
* Hyperoxaluria or history of nephrolithiasis
* Left ventricular ejection fraction < 40%
* Contraindications to beta-blocker or vitamin C.
* Patients with history of vitamin C consumption before surgery.
* Chronic kidney disease with creatinine >2 mg/dl.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative atrial fibrillation (POAF) incidence in patients undergoing coronary artery bypass (CABG) surgery through the administration of vitamin C supplementation compared to placebo group | through hospital stay , an average of 7 days
  Evaluate the effectiveness of perioperative oral vitamin C in prevention for post operative AF following elective on-pump coronary artery bypass surgery in old adult Egyptian.
  patients during hospital stay.
compare between high dose verses low dose of vitaminC | through hospital stay, an average of 7 days
  Quantify the effective dose of perioperative oral vitamin C on the incidence of the POAF during hospital stay following elective on-pump CABG surgery in old adult Egyptian patients.

SECONDARY OUTCOMES:
Lenght of hospital stay | through hospital stay, an average of 7 days
  Estimate the impact of of perioperative oral vitamin C supplementation on hospital length of stay following elective on-pump CABG surgery in old adult Egyptian patients.

CONTACTS AND LOCATIONS:
Locations (1):
- El Sheik Zayed Specialized Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No